CLINICAL TRIAL: NCT04084418
Title: Carbohydrates Under Target for Type 1 Diabetes Management
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lock down due to COVID-19 pandemic.
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Anne-Sophie Brazeau, Assistant Professor, McGill University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CUT-T1D
Record Dates: First submitted 2019-09-04; First posted 2019-09-10 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control diet followed by VLCHF diet (Experimental): * Phase 1 (1 to 3 weeks): Insulin dose optimization with usual diet
  * Phase 2 (6 weeks): Control diet (50% of energy from carbohydrates)
  * Phase 3 (4 weeks): Washout period
  * Phase 4 (6 weeks): VLCHF diet (10% of energy from carbohydrates)
  Interventions: Other: Control Diet; Other: VLCHF Diet
- VLCHF diet followed by Control diet (Experimental): * Phase 1 (1 to 3 weeks): Insulin dose optimization with usual diet
  * Phase 2 (6 weeks): VLCHF diet (10% of energy from carbohydrates)
  * Phase 3 (4 weeks): Washout period
  * Phase 4 (6 weeks): Control diet (50% of energy from carbohydrates)
  Interventions: Other: Control Diet; Other: VLCHF Diet

INTERVENTIONS:
Other: Control Diet — Participants will be provided with a two-week menu to be consumed 3 times for each intervention, for a total of 6 weeks per intervention. For the Control diet, the diet will provide 50% of energy from CHO, 15% from protein, and 35% from lipids. Menu will be adapted to the participant's food preferences and usual caloric intake by a dietitian. Participants will be asked to limit their alcohol intake in both interventions. During this phase, participants will also have to wear a pedometer and use the Pezio: Achieve the Guidelines! mobile application to help the research assistant track their daily steps remotely.
Other: VLCHF Diet — Participants will be provided with a two-week menu to be consumed 3 times for each intervention, for a total of 6 weeks per intervention. For the Experimental diet, the diet will provide 10% of energy from CHO, 15% from protein, and 75% from lipids. During the Experimental diet, participants will be provided with a multivitamin to reduce risk of deficiencies due to restrictions on fruits and grain products. Menu will be adapted to the participant's food preferences and usual caloric intake by a dietitian. Participants will be asked to limit their alcohol intake in both interventions. During this phase, participants will also have to wear a pedometer and use the Pezio: Achieve the Guidelines! mobile application to help the research assistant track their daily steps remotely.

SUMMARY:
Recently there has been an increased interest in limiting intake of carbohydrates (CHO) for improving long term health. While healthcare professionals (HCPs) are sometimes reluctant to limit the CHO intake due to the lack of information related to safety issues, low CHO diets are increasing in popularity amongst both people with and without diabetes. One of these diets, the very low CHO high fat diet (VLCHF) raises concern on its impact on the lipid profile, liver, response to glucagon, and insulin dose adjustments when adopting it in the context of type 1 diabetes (T1D). The investigators recently conducted a series of interviews with people with diabetes following a VLCHF diet (Brazeau et al. Manuscript in preparation) to inquire on their reasons for adopting VLCHF as well as challenges they faced. The main reasons to initiate the diet were to limit blood glucose fluctuations and reduce medication. An issue that was frequently mentioned during the interviews was the lack of support from HCPs which often leads to not discussing it with said HCP. This is an important source of concern that can lead to additional safety issues. Our goal is to provide information regarding the safety of a VLCHF diet for T1D and the individualized insulin adjustments required.

The investigators aim to evaluate the changes in daily blood glucose fluctuations after 6 weeks of a VLCHF diet, to monitor the changes in the insulin dosing and to measure impact on lipid profiles, response to glucagon, and liver function.

ELIGIBILITY:
Inclusion Criteria:

* Duration of Type 1 Diabetes > 12 months
* On intensive insulin therapy for > 6 months
* Own a smartphone or tablet to use two mobile applications : Keenoa and Piezo: Achieve the Guidelines!

Exclusion Criteria:

* Known gastroparesis (clinical diagnosis)
* Advanced kidney disease (eGFR < 50 mL/min)
* Known significant liver disease (e.g., cirrhosis, active hepatitis, liver transplantation)
* Recent (< 6 months) major cardiovascular even (e.g. myocardial infarction, cerebrovascular accident, major revascularization, etc.)
* Pregnancy (ongoing or planned in the next 6 months)
* Breastfeeding
* Severe hypoglycemia episodes or ketoacidosis in the 4 weeks prior to recruitment
* Claustrophobia or presence of metal devices/implants in the body

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2020-03-23 (Actual); Study Completion 2020-03-23 (Actual)

PRIMARY OUTCOMES:
Daily blood glucose standard deviation | Over the 6 weeks of each intervention diet
  Using continuous glucose monitoring

SECONDARY OUTCOMES:
Percentage of time-in-target (range of 4-10 mmol/L) | Over the 6 weeks of each intervention diet
  Using continuous glucose monitoring
Coefficient of glucose variation | Over the 6 weeks of each intervention diet
  Using continuous glucose monitoring
Mean sensor glucose values (mmol/L) | Over the 6 weeks of each intervention diet
  Using continuous glucose monitoring
Glucose area under the curve for 2 hours post-prandial | First and last week of each intervention diet
  Using continuous glucose monitoring
Number of hypoglycemia episodes necessitating treatment recorded | Over the 6 weeks of each intervention diet
  Recorded by participants on hypoglycemia journal
Percentage of time spent in hypoglycemia ranges (< 4 mmol/L and < 3 mmol/L) | Over the 6 weeks of each intervention diet
  Using continuous glucose monitoring
Percentage of time spent in hyperglycemia ranges (>10 mmol/L and > 15 mmol/L) | Over the 6 weeks of each intervention diet
  Using continuous glucose monitoring
Daily insulin adjustments required to maintain safe blood glucose | Over the 6 weeks of each intervention diet
  Adjustments (basal and prandial) to avoid hypoglycemia (blood glucose < 4 mmol/L) and hyperglycemia (blood glucose > 15 mmol/L)
Short-term effects on anthropometric parameters : weight (kg) and height (cm) | Following the 6 weeks of each intervention diet
  Weight and height will be combined to report BMI (kg/m^2)
Short-term effects on anthropometric parameters : waist circumference (cm) | Following the 6 weeks of each intervention diet
  Calculated using the average of 3 measures
Short-term effects on blood lipid profiles | Following the 6 weeks of each intervention diet
  Total cholesterol, HDL-chol, and LDL-chol, triglycerides, Apo-B and Apo-A
Short-term effects on body composition (lean and fat mass) | Following the 6 weeks of each intervention diet
  Measured by DEXA (Dual-Energy X-ray Absorptiometry)
Short-term effects on inflammatory parameters | Following the 6 weeks of each intervention diet
  Plasma lipopolysaccharide (LPS), interleukine 6 (IL-6), monocyte chemoattractant protein-1 MCP-1)
Short-term effects on oxidative stress/redox parameters | Following the 6 weeks of each intervention diet
  Total and reduced glutathione
Short-term effects on blood pressure | Following the 6 weeks of each intervention diet
  Systolic and diastolic blood pressure
Short-term effects on liver function | Following the 6 weeks of each intervention diet
  Aminotransferases, alkaline phosphatase, gamma-glutamyl transpeptidase, bilirubin, albumin
Short-term effects on resting metabolic rate | Following the 6 weeks of each intervention diet
  After a 10-hour fast measured by indirect calorimetry
Short-term effects on liver proton density fat fraction by MRS (MRS-PDFF) (%) | Following the 6 weeks of each intervention diet
  Using hepatic fat imagery (MRI)
Short-term effects on mean liver PDFF | Following the 6 weeks of each intervention diet
  Using hepatic fat imagery (MRI)
Short-term effects on total liver volume (mL) | Following the 6 weeks of each intervention diet
  Using hepatic fat imagery (MRI)
Short-term effects on total liver fat index (%.ml) | Following the 6 weeks of each intervention diet
  Using hepatic fat imagery (MRI)
Efficacy of glucagon in correcting hypoglycemia | Following the 6 weeks of each intervention diet
  Time needed to reach a blood glucose > 4 mmol/L after glucagon treatment of an insulin-induced hypoglycemia reaching 4 mmol/L at 15, 20 and 30 min post glucagon administration, peak plasma glucose level two hours after administration, insulin, glucagon, ketone and free fatty acids levels.
Modulation of postprandial glycemic response (Standardized meal-tests) | Following the 6 weeks of each intervention diet
  Hunger, appetite and fullness scores, lat the following times (-20, 0, 15, 30, 60, 90, 120 and 180 min, with 0 min being the start of meal consumption)
Secretion of key gastrointestinal peptides (Standardized meal-tests) | Following the 6 weeks of each intervention diet
  Gastrointestinal peptides : levels of glucose, insulin glucagon, GLP-1, PYY and acylated ghrelin at the following times (-20, 0, 15, 30, 60, 90, 120 and 180 min, with 0 min being the start of meal consumption), as well as their corresponding kinetics including areas under the curve (AUC), peak values and nadirs.
Questionnaire of well-being (score) | Following the 6 weeks of each intervention diet
  Corresponding scores of questionnaire used to assess different quality of life aspects: well-being, fatigue, nausea, hunger, appetite, desire to eat.
Questionnaire of diet satisfaction (score) | Following the 6 weeks of each intervention diet
  Corresponding scores of questionnaire used to assess different quality of life aspects: diet satisfaction, difficulty to follow the diet, difficulty for meal preparation.
Effects on physical activity (steps/day) | Over the 6 weeks of each intervention diet
  Steps per day recorded with a pedometer (PedioRxD) and mobile application (baseline and during each intervention diet)

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de recherches cliniques de Montréal, Montreal, Quebec, Canada